CLINICAL TRIAL: NCT04323852
Title: Vitamin D Treatment Attenuates Heart Apoptosis After Coronary Artery Bypass Surgery; A Double-Blind Randomized Placebo-Controlled Clinical Trial
Brief Title: Can Vitamin D Reduce Heart Muscle Damage After Bypass Surgery?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Erfan Tasdighi, Principle investigator, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 13312; ISRCTN44896820 (Registry Identifier: ISRCTN); IRCT20180118038423N1 (Registry Identifier: IRCT)
Record Dates: First submitted 2020-03-23; First posted 2020-03-27 (Actual); Results first posted 2021-10-19 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-09

CONDITIONS: Vitamin D Deficiency; Cardiomyopathies; Apoptosis; Inflammation
Keywords: Vitamin D; Cardiovascular disease; Apoptosis; Insulin-like growth factor-1; Coronary artery disease; Cardiopulmonary bypass; Interleukin-10
MeSH Terms: conditions — Vitamin D Deficiency; Cardiomyopathies; Inflammation; Cardiovascular Diseases; Coronary Artery Disease | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: With the exception of the pharmacists, all the investigators, patients and the medical team were blinded to the group allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- vitamin D (Experimental): 35 patients that pass the inclusion criteria and do not have exclusion criteria that will receive Vitamin D for 3 days and each time 3 doses of 50000 units
  Interventions: Drug: Vitamin D
- control group (Placebo Comparator): 35 patients that will receive placebo for 3 days and each day for 3 doses
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin D — Participants undergoing coronary artery bypass graft (CABG) surgery are randomly allocated to group A (intervention), who receive 3 doses of vitamin D (50000 U) a day for 3 days before surgery
  Arms: vitamin D
Drug: Placebo — Placebo
  Arms: control group

SUMMARY:
Background and study aim:

Heart diseases are among the most common causes of death worldwide. A large proportion of deaths are caused by heart attacks (myocardial infarction), where blood flow to the heart is reduced resulting in damage to the heart muscle. If the arteries supplying blood to the heart start to become blocked, Coronary Artery Bypass Grafting (CABG) surgery is a treatment to replace the blocked sections of artery can reduce angina (chest pain). However, CABG surgery has complications, including an increased risk of heart attack. Vitamin D deficiency is thought to be linked to poorer recovery from heart attack and CABG surgery. This study aims to investigate if vitamin D supplementation can reduce injury to the heart following CABG surgery.

Who can participate? Adults with vitamin D deficiency undergoing CABG

What does the study involve? Participants are randomly allocated to one of two groups. Those in the first group receive vitamin D at 3 doses per day for 3 days before surgery. The second group will receive a dummy pill (placebo). Both groups will have standard CABG surgery.

What are the possible benefits and risks of participating? Those in the vitamin D group might benefit from its effects. Vitamin D has few side effects, especially when taken for only a few days.

Where is the study run from? Shahid Modarres Hospital (Iran)

When is the study starting and how long is it expected to run for? September 2017 to January 2019

Who is funding the study? Deputy of Research of Shahid Beheshti School of Medicine

Who is the main contact? Dr Erfan Tasdighi erfan.tasdighi@gmail.com

DETAILED DESCRIPTION:
Enrollment started in June 2018 and was completed in December 2018. The inclusion criteria were as following: the patients referred for elective and isolated Coronary Artery Bypass Graft (CABG) using Cardiopulmonary Bypass (CPB) with vitamin D deficiency (defined as 25-hydroxyvitamin D [25(OH) D] < 20 ng/mL) and normal kidney function (creatinine <1.5mg/dL). The exclusion criteria were: recent myocardial infarction, urgent CABG, non-isolated coronary surgery, redo surgery, malignant disease, presence of acute or chronic inflammatory diseases, history of vitamin D treatment within previous 6 months, or unwillingness to participate.

Intervention Following informed consent, eligible study participants were randomly assigned (by using a computer- generated random code) in a 1:1 ratio to receive either placebo or a total of 450,000 international units (IU) vitamin D3 (three 50,000 IU of vitamin D3 tablet daily for 3 days) before operation. The placebo group received three inactive medication tablets daily at the same time point. With the exception of the pharmacists, all the investigators, patients and the medical team were blinded to the group allocation.

Coronary artery bypass was done in the culprit lesions for both groups by one surgical team. The standard protocol for general anesthesia, surgical and CPB management were performed for all patients and have already been described in detail [16].

Outcome measures The primary outcome was the degree of heart apoptosis by measurement of caspase 2, 3 and 7 activity from right atrial specimen with immunohistochemistry staining, and the serum level of anti-inflammatory interleukin-10 (IL-10) and insulin- like growth factor (IGF-1), and N-terminal pro v-type Brain Natriuretic Peptide (nt-pro BNP). The biopsy from right atrial appendage was taken at the end of surgery after venous cannula removal in a nontraumatic fashion, kept into formalin and in less than 24h parafinized. Blood samples were collected at the baseline (T1), before anesthesia induction (T2), at the end of surgery after protamine reversal (T3) and the first postoperative day (T4) to measure the serum level of IGF-1, IL-10 and pro BNP. The blood samples were centrifuged at 2500 rpm for 15 min within one hour after blood sampling, and the serum was stored at -20°C until assayed.

Enzyme-linked immunosorbent assay The concentration of IL-10 was measured by a quantitative ELISA kit . The concentration of the IGF- 1 was measured by a quantitative ELISA kit .

Serum vitamin D was detected by using the high performance liquid chromatography method . The pro BNP measurement was done using a commercially available two- site chemiluminescent immunometric assay .

Immunohistochemistry studies Immunohistochemical staining was performed on 5-micrometer thick sections. The slides were incubated at 37°C for 24 hours and de-paraffinized in pre-heated xylene and rehydrated through descending grades of alcohol, washed in distilled water. Heat induced antigen retrieval was done by microwave oven with citrate buffer (pH 6.0) for anti-caspase-7 and Ethylenediamine Tetraacetic Acid; buffered solution (Tris-EDTA) (pH=8) for anti-caspase-2 and 3. endoperoxidase blocking was done by adding hydrogen peroxide on the sections. The protein block then added for 5 minutes, slides were washed in Tris-Buffered Saline (TBS). .The primary antibody as anti-caspase-2 antibody, rabbit monoclonal , anti-caspase-3 antibody, rabbit monoclonal , anti-caspase-7 antibody, and mouse monoclonal (clone 7-1-11 , abcam) antibody were added and kept for 30 minutes, washed in TBS. Mouse and Rabbit Specific horseradish peroxidase/Diaminobenzidine (HRP/DAB) immunohistochemistry (IHC) Detection Micro-polymer Kit were used and incubated for 15 minutes then washed with tris-buffered saline (TBS). Diaminobenzidine (DAB) chromogen was added and kept for 5 minutes. Slides washed in distilled water and counter stained with hematoxylin. Sections containing lymph node tissue were used as positive control. Negative control included primary antibody replaced with phosphate buffered saline (PBS). Immunostained sections were reviewed for cytoplasmic expression of anti-caspase-2, anti-caspase-3 and anti-caspase-7. The number of immune-reactive cells per High Power Field (HPF) (X 400) was counted. For this purpose at least 10 HPF were assessed and the average of positive cells was recorded.

Sample size and statistical methods The determination of the patient number (30 patients per group) was based on previous trials investigating the caspase activity in the CABG setting .

Categorical variables were reported as numbers and percentages, whereas mean± standard deviation was expressed for continuous variables. Repeated measures of analysis of variance and multiple comparisons using the Bonferroni correction (type I error correction) were applied for evaluating the change of measured inflammatory markers between the groups over time. The Kolmogorov-Smirnov test for normality was performed. Continuous variables and categorical variables were compared between groups using Student's t test (or Mann-Whitney test for those meeting abnormal distribution) and Chi-square, respectively. All the statistical analyses were performed using SPSS version 23 (SPSS, Chicago, IL, USA). A p values <0.05 was considered to be significant.

ELIGIBILITY:
Inclusion Criteria:

1. Candidate for first-time elective CABG surgery for coronary artery disease (CAD)
2. Coronary artery surgery only (i.e. no valvular surgery)
3. Cardiopulmonary pump used during surgery
4. Vitamin D level below 30 ng/ml

Exclusion Criteria:

1. Renal failure or creatinine level >1.5 mg/dl
2. Previous use of vitamin D supplement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-01-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erfan Tasdighi, MD, Principal Investigator — Shahid Beheshti university of medical science
Locations (1):
- modarres Hospital, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vitamin D | Control Group
Started | 35 | 35
Completed | 35 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin D | Control Group | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (6) | 58 (9) | 58.5 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 27 | 28 | 55
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Iran | 35 | 35 | 70
Ejection Fraction [Mean (Standard Deviation); unit: percentage] | 47 (10) | 48 (9) | 47.5 (8)
Myocardial infarction [Count of Participants; unit: Participants] | 19 | 15 | 34
Erythrocyte sedimentation rate (ESR) [Mean (Standard Deviation); unit: mm/hour] | 13 (9) | 14 (8) | 13.6 (4)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27 (3) | 27 (3) | 27 (1)
25 (OH)D [Mean (Standard Deviation); unit: ng/mL] | 12.8 (6) | 12.1 (5) | 12.4 (4)
Hyperlipidemia [Count of Participants; unit: Participants] | 9 | 16 | 25
Diabetes Mellitus [Count of Participants; unit: Participants] | 12 | 19 | 31
Hypertension [Count of Participants; unit: Participants] | 18 | 22 | 40
Smokers [Count of Participants; unit: Participants] | 15 | 21 | 36
Family history of cardiovascular disease [Count of Participants; unit: Participants] | 9 | 8 | 17

OUTCOME MEASURES:

1. Primary Outcome: Caspase 2 Enzyme Level
Description: Caspase 2 enzyme activity in right atrial specimen measured by with immunohistochemistry staining The positive control and negative control were taken from human lymph node tissue. as for the control tissue a humane lymph node was used. Positivity for active caspase is shown using cytoplasmic staining . the number of apoptotic cells was measure per each high power filed (HPF) under light microscopy.
Time Frame: during the surgery, an average of 3 hours
Measure: Mean (Standard Deviation); unit: cells/ HPF
Arm/Group | Vitamin D | Control Group
Number analyzed (Participants) | 35 | 35
cells/ HPF | 1.3 (1.0) | 2.0 (0.9)

2. Primary Outcome: Caspase 3 Enzyme Level, an Average of 3 Hours
Description: Caspase 3 enzyme activity in right atrial specimen measured by with immunohistochemistry staining The positive control and negative control were taken from human lymph node tissue. as for the control tissue a humane lymph node was used. Positivity for active caspase is shown using cytoplasmic staining . the number of apoptotic cells was measure per each high power filed (HPF) under light microscopy.
Time Frame: during the surgery, an average of 3 hours
Measure: Mean (Standard Deviation); unit: cells/ HPF
Arm/Group | Vitamin D | Control Group
Number analyzed (Participants) | 35 | 35
cells/ HPF | 1.2 (0.8) | 2.0 (0.8)

3. Primary Outcome: Caspase 7 Enzyme Level
Description: Caspase 7 enzyme activity in right atrial specimen measured by with immunohistochemistry staining The positive control and negative control were taken from human lymph node tissue. as for the control tissue a humane lymph node was used. Positivity for active caspase is shown using cytoplasmic staining . the number of apoptotic cells was measure per each high power filed (HPF) under light microscopy.
Time Frame: during the surgery, an average of 3 hours
Measure: Mean (Standard Deviation); unit: cells/ HPF
Arm/Group | Vitamin D | Control Group
Number analyzed (Participants) | 35 | 35
cells/ HPF | 1.3 (1.0) | 1.8 (1.2)

4. Primary Outcome: Interlukin-10 (IL-10) Serum Level
Description: The concentration of IL-10 in the serum of patients was measured using a quantitative enzyme-linked immunosorbent assay (ELISA) kit .
Time Frame: Right before the intervention(3 days before surgery)
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Vitamin D | Control Group
Number analyzed (Participants) | 35 | 35
pg/ml | 1.0 (0.35) | 1.0 (0)

5. Primary Outcome: Interleukin-10 (IL-10) Serum Level
Description: as for outcome 4
Time Frame: procedure (before anesthesia induction)
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Vitamin D | Control Group
Number analyzed (Participants) | 35 | 35
pg/ml | 4.4 (4.9) | 1.0 (0)

6. Primary Outcome: Interleukin--10 (IL-10) Serum Level
Description: as for outcome 4
Time Frame: at the end of surgery after protamine reversal
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Vitamin D | Control Group
Number analyzed (Participants) | 35 | 35
pg/ml | 304.8 (85.6) | 205.5 (107.4)

7. Primary Outcome: Interleukin (IL-10) Serum Level
Description: as for outcome 4
Time Frame: the first postoperative day
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Vitamin D | Control Group
Number analyzed (Participants) | 35 | 35
pg/ml | 7.6 (6.5) | 4.0 (6.7)

8. Primary Outcome: Insulin Growth Factor
Description: The concentration of the IGF-1 was also measured by a quantitative ELISA kit
Time Frame: Right before the intervention(3 days before surgery)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Vitamin D | Control Group
Number analyzed (Participants) | 35 | 35
ng/mL | 86.3 (33.9) | 76.5 (26.6)

9. Primary Outcome: Insulin Growth Factor
Description: The concentration of the IGF-1 was also measured by a quantitative ELISA kit
Time Frame: procedure (before anesthesia induction)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Vitamin D | Control Group
Number analyzed (Participants) | 35 | 35
ng/mL | 109.8 (63.2) | 75.0 (21.3)

10. Primary Outcome: Insulin Growth Factor
Description: The concentration of the IGF-1 was also measured by a quantitative ELISA kit
Time Frame: at the end of surgery after protamine reversal
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Vitamin D | Control Group
Number analyzed (Participants) | 35 | 35
ng/mL | 142.0 (67.1) | 82.1 (35.9)

11. Primary Outcome: Insulin Growth Factor
Description: The concentration of the IGF-1 was also measured by a quantitative ELISA kit
Time Frame: the first postoperative day
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Vitamin D | Control Group
Number analyzed (Participants) | 35 | 35
ng/mL | 108.6 (61.2) | 69.4 (35.4)

12. Secondary Outcome: Hemorrhage After Surgery
Description: after the surgery all the hemorrhage of patients was collected by suctioning and the exact amount of bleeding has been reported.
Time Frame: immediately after surgery
Measure: Mean (Standard Deviation); unit: cc
Arm/Group | Vitamin D | Control Group
Number analyzed (Participants) | 35 | 35
cc | 360.7 (237.7) | 404.4 (245.9)

13. Secondary Outcome: Blood Units Usage
Description: number of pack cell that was administered for the patient
Time Frame: discharge 1 day
Measure: Mean (Standard Deviation); unit: units
Arm/Group | Vitamin D | Control Group
Number analyzed (Participants) | 35 | 35
units | 0.5 (0.7) | 0.8 (0.9)

14. Secondary Outcome: Ventilator Application
Description: period of time that the patient was on ventilator
Time Frame: discharge 1 day
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Vitamin D | Control Group
Number analyzed (Participants) | 35 | 35
hr | 6.8 (2.3) | 8.3 (4.4)

15. Secondary Outcome: Creatinine Level
Description: The serum level of Creatinine in the patients which is a measurement of the kidney function
Time Frame: immediately after surgery
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Vitamin D | Control Group
Number analyzed (Participants) | 35 | 35
mg/dl | .8 (.05) | .9 (.04)

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Vitamin D | Control Group
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 4/35 | 5/35
Other Adverse Events (participants affected / at risk) | 7/35 | 7/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitamin D (N=35) | Control Group (N=35)
brain stroke (Nervous system disorders) | 2 (3) | 2 (2) — A stroke occurs when the blood supply to part of your brain is interrupted or reduced, preventing brain tissue from getting oxygen and nutrients
heart attack (Cardiac disorders) | 1 (1) | 2 (2) — A heart attack happens when the flow of oxygen-rich blood in one or more of the coronary arteries, which supply the heart muscle, suddenly becomes blocked, and a section of heart muscle can't get enough oxygen
gastrointestinal bleeding (Gastrointestinal disorders) | 1 (2) | 1 (2) — Gastrointestinal (GI) bleeding is a symptom of a disorder in your digestive tract. The blood often appears in stool or vomit but isn't always visible, though it may cause the stool to look black or tarry
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitamin D (N=35) | Control Group (N=35)
DVT (Vascular disorders) | 2 (3) | 1 (2) — Deep vein thrombosis (DVT) is a medical condition that occurs when a blood clot forms in a deep vein
infection (Immune system disorders) | 5 (6) | 6 (7) — The invasion and growth of germs in the body

LIMITATIONS AND CAVEATS:
Although this single-center study had a relatively small sample size and was limited to cardiac surgery patients, the study design was RCT with homogenous patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-10-24): https://cdn.clinicaltrials.gov/large-docs/52/NCT04323852/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-24): https://cdn.clinicaltrials.gov/large-docs/52/NCT04323852/SAP_001.pdf